CLINICAL TRIAL: NCT05250076
Title: Immediate Effects of Kinesio Tape on Median Nerve's Mechanosensitivity, Measured by the Upper Limb Neurodynamic Test 1 (ULNT1) in Healthy Participants: A Randomized Controlled Trial
Brief Title: Immediate Effects of Kinesio Tape on Median Nerve's Mechanosensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FISIO-2-28102019
Record Dates: First submitted 2022-01-13; First posted 2022-02-22 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): The beige Kinesio Tape (Prim Tape®) will be applied, from distal to proximal, 5cm wide, cut in "I" and with tension below 50%. The Kinesio Tape will be placed along the entire path of the median nerve, from the wrist to the armpit. The participants will remain in the supine position on a treatment table (Posturarte® Olympic), without inclination (Posturarte® Olympic). To clean the participant's skin, cotton (MASMI®) will be passed with ethyl alcohol (Fergus®). Scissor (Maped®) will be used to cut the Kinesio Tape.
  Interventions: Device: Kinesio Tape
- Control Group (No Intervention): The participants will remain at rest in a supine position on a treatment table (Posturarte® Olympic) without inclination for 5 minutes.

INTERVENTIONS:
Device: Kinesio Tape — The beige Kinesio Tape (Prim Tape®) will be applied, from distal to proximal, 5cm wide, cut in "I" and with tension below 50%. The Kinesio Tape will be placed along the entire path of the median nerve, from the wrist to the armpit. The participants will remain in the supine position on a treatment table (Posturarte® Olympic), without inclination.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to verify the immediate effects of Kinesio Tape on median nerve's mechanosensitivity, measured by the upper limb neurodynamic test 1 (ULNT1) in healthy participants.

DETAILED DESCRIPTION:
After completing the socio-demographic and clinical questionnaire, the participants will be randomly assigned into two designated groups, the Intervention Group (IG; n = 30) (Kinesio tape throughout the median nerve course) and the Control Group (CG; n = 30) (remained at rest for 5 minutes), using the software www.graphpad.com/quickcals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students of both genders with normal mobility of the joints of the upper quadrant of the body

Exclusion Criteria:

* Deformities in the upper quadrant region of the body;

  * Complaints in this region in the last 6 months;
  * Surgical procedures or musculoskeletal, cardiac, renal, metabolic, neurological and or oncological pathologies of the upper quadrant that may disturb nerve function;
  * Not present any mechanosensitive response to ULNT1;
  * Pregnant women;
  * Ingestion of non-steroidal anti-inflammatory drugs or consumption of any type of narcotic drugs and participants who have drunk alcohol in the last 12 hours.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-03-26 (Actual)

PRIMARY OUTCOMES:
change in elbow extension range of motion measured by smartphone | [Time Frame: Baseline (Moment 0), Immediately after intervention or control (Moment 1) .]]
  Data will be collected in two moments: baseline (Moment 0) and after the application of Kinesio Tape for intervention group or after a resting period for control group (Moment 1).
  Moment 0 will consist in performing the ULNT1 on the dominant upper limb for each participant. The participants will remain in a supine position on a treatment table with the body aligned, exposing the test forearm for the placement of the smartphone through an armband. The head and cervical spine will be stabilized at the maximum comfortable lateral inclination using a foam pillow. The ULNT1 sequence used was: (1) maximum contralateral cervical inclination; (2) arm at 90º of shoulder abduction preventing scapular elevation; (3) 90º of external rotation of the shoulder and elbow flexion at 90º (defined as the initial position or 0º of range of motion under test); (4) supination of the forearm; (5) wrist and fingers extension; and (6) elbow extension.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cardoso, PhD, Principal Investigator — Fernando Pessoa University
Locations (1):
- Ricardo Cardoso, Porto, Portugal